CLINICAL TRIAL: NCT04261738
Title: Effects of Hyperbaric Oxygen Therapy on Glucose Homeostasis in Patients Living With Diabetes Mellitus
Brief Title: Effects of HBO on Glucose in Patients With DM
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Facility closure, awaiting relocation
Sponsor: Legacy Health System (Other)
Collaborators: DexCom, Inc. (Industry)
Responsible Party: Principal Investigator, Enoch Huang, Medical Director, Hyperbaric Medicine and Wound Care Clinic, Legacy Health System
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HB-002
Record Dates: First submitted 2020-02-06; First posted 2020-02-10 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1
Keywords: hyperbaric oxygen; continuous glucose monitor; hbo; cgm
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus, Type 1 | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Intervention Model Description: Control exposure followed by Hyperbaric Oxygen exposure
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Control (No Intervention): The first 2-hour session will be a control where participants will sit quietly (as they would in the hyperbaric chamber) and will not be allowed to consume carbohydrates unless directed to by the hyperbaric department hypoglycemia protocol.
- Hyperbaric Oxygen (Experimental): The following day for the HBO2 session, subjects will be fitted for an oxygen hood and given a standard HBO2 treatment. In the chamber the pressure will increase to approximately 2-1/2 times normal atmospheric pressure (2.4 atmospheres absolute [ATA]). Once they reach the treatment pressure, subjects will breathe oxygen by placing the hood over their head and securing it in place. They will breathe oxygen for a 30-minute period, and then take the hood off for 5 minutes for an "air break." They will have a total of three 30-minute oxygen periods and two 5-minute air breaks. A subject will be in the hyperbaric chamber for approximately 2 hours.
  Interventions: Device: Hyperbaric Oxygen

INTERVENTIONS:
Device: Hyperbaric Oxygen — Volunteers will be given a standard hyperbaric oxygen treatment (2.4 ATA x 90 minutes)
  Other Names: HBOT; HBO2
  Arms: Hyperbaric Oxygen

SUMMARY:
The purpose of this Research Study is:

1. To determine the reliability and performance of the Dexcom G6® continuous glucose monitoring (CGM) system in patients with diabetes undergoing hyperbaric oxygen (HBO2) exposure. The study-specific blood glucose meter and CGM system are approved by the FDA (U.S. Food and Drug Administration).
2. To determine whether HBO2 exposure causes blood glucose to drop as a result of the treatment.
3. To determine whether HBO2 causes a change in blood glucagon (a hormone that raises blood glucose).

Investigators will be comparing changes in blood glucose and glucagon in volunteers with diabetes who will be exposed to a single hyperbaric oxygen treatment (pressurization to 2.4 atmospheres absolute for 90 minutes) to a control period of 2 hours where volunteers will simulate a hyperbaric treatment while sitting in an examination room breathing room air at sea level pressure. Investigators will be measuring blood glucose with a variety of devices including a continuous glucose monitor, two point-of-care glucometers, and the hospital inpatient laboratory measurement of venous blood.

DETAILED DESCRIPTION:
The purpose of this Research Study is to determine whether the Dexcom G6® continuous glucose monitoring (CGM) system accurately estimates blood glucose in diabetic patients undergoing hyperbaric oxygen (HBO2) exposure. The study-specific CGM system is approved by the FDA (U.S. Food and Drug Administration).

Subjects will have the Dexcom CGM inserted underneath the skin of their abdomen. This is done in the office. It is secured to the skin by use of an adhesive patch. The sensor measures glucose levels just underneath the skin. A transmitter is fastened on top of the sensor and sends this information wirelessly to a receiver or compatible smart device. Study participants will also have second sensor inserted in the subcutaneous tissue on the back of the arm as a backup in case of data loss. The subjects will wear the sensors for at least 48 hours and then return to the Hyperbaric Medicine Clinic.

At the Hyperbaric Medicine Clinic, study staff will check the CGM system to make sure it has been working properly. The first 2-hour session will be a control where participants will sit quietly (as they would in the hyperbaric chamber) and will not be allowed to consume carbohydrates unless directed to by the hyperbaric department hypoglycemia protocol. The following day for the HBO2 session, subjects will be fitted for an oxygen hood and given a standard HBO2 treatment. Investigators will obtain concurrent transcutaneous oximetry measurements (TCOM) attached no farther than 3 cm from the commercial CGM on the abdomen to measure tissue oxygenation in the region of the CGM only during HBO2 exposure.

The hyperbaric oxygen therapy chamber can accommodate 12 patients at a time. Study subjects could be in the chamber along with regularly scheduled patients. In the chamber the pressure will increase to approximately 2-1/2 times normal atmospheric pressure (2.4 atmospheres absolute [ATA]). Once they reach the treatment pressure, subjects will breathe oxygen by placing the hood over their head and securing it in place. They will breathe oxygen for a 30-minute period, and then take the hood off for 5 minutes for an "air break." They will have a total of three 30-minute oxygen periods and two 5-minute air breaks. A subject will be in the hyperbaric chamber for approximately 2 hours.

Blood sampling will be identical for both the control and HBO2 exposure days. Subjects will have a peripheral intravenous (IV) catheter placed and a total of 12 samples collected to measure venous blood glucose (12 timepoints), glucagon levels (3 timepoints) and HgA1c, (one time). A RN or MD will be inside the chamber to monitor the subjects and to obtain the IV blood samples. Because CGMs have not been established to be reliable under HBO2 conditions in patients with DM, the protocol will collect Point-of-Care (POC) glucose measurements using the hospital's standard glucometer (Nova Biomedical, Waltham, MA) and the AccuChek Inform II POC glucometer (Roche Diagnostics, Indianapolis, IN) at each testing point. This will be done using a lancet to pierce the skin of the fingertip to get a drop of blood.

Subjects in both groups will also be required to perform home glucose monitoring (4 times per day) and record mealtimes and the time of any medications taken throughout the study period.

Subjects will return to the clinic on Day 10. The CGM sensor will be removed and the transmitter and display device collected by staff. Removed sensors will be returned to the manufacturer for analysis. That is the end of the subject's study participation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 1 or type 2 diabetes
* Willing to have 2 subcutaneous glucose monitors for 10 days
* Willing to be NPO after midnight on the day of the study session
* Willing to come to the hyperbaric facility on successive days (one control session and one hyperbaric treatment), spending approximately 3 hours in the facility on each day of testing
* Willing to undergo multiple fingersticks on the days of testing
* Willing to have a peripheral intravenous catheter placed for blood sampling
* Willing to perform four daily fingerstick blood glucose checks throughout the study period

Exclusion Criteria:

* Contraindication to HBO2 as determined by the study investigator (e.g., pregnancy)
* Previous treatment with HBO2 within 30 days of enrollment
* Current use of CGM is not an exclusion, but participants must use study equipment during the study
* Current use of an insulin pump
* Known allergy to medical-grade adhesives
* Extensive skin changes/disease that preclude wearing the sensor on normal skin (e.g. extensive psoriasis, recent burns or severe sunburn, extensive eczema, extensive scarring, extensive tattoos, dermatitis herpetiformis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-09-02 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
CGM Reading | 10 days
  Estimated glucose value from the continuous glucose monitor
CGM Reading from Data Logger | 10 days
  Estimated glucose value from the data logger
Fingerstick point of care glucose | 2 days
  Estimated glucose value from fingersticks during control and HBOT arms
Fingerstick point of care glucose | 10 days
  Estimated glucose value from fingersticks during the length of the study (4 times/day)
Hospital laboratory glucose | 2 days
  Estimated glucose value from venous blood during control and HBOT arms
Hba1c | One time only on day 3 of study
  Baseline Hba1c

SECONDARY OUTCOMES:
Glucagon | 2 days
  We will determine whether HBOT has any effect on glucagon levels on control and HBOT arm

CONTACTS AND LOCATIONS:
Overall Officials: Enoch Huang, MD, Principal Investigator — Legacy Emanuel Medical Center
Locations (1):
- Legacy Emanuel Medical Center, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Huang E, Demirel S, Bliss C, Savaser D, Castle JR. Reliability of the Dexcom G6 Continuous Glucose Monitor During Hyperbaric Oxygen Exposure. Diabetes Technol Ther. 2020 May;22(5):360-366. doi: 10.1089/dia.2019.0390. Epub 2020 Feb 6. PMID 31916854

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-12-04): https://cdn.clinicaltrials.gov/large-docs/38/NCT04261738/Prot_SAP_001.pdf
  • Informed Consent Form (2019-12-17): https://cdn.clinicaltrials.gov/large-docs/38/NCT04261738/ICF_000.pdf